CLINICAL TRIAL: NCT03094299
Title: The Efficacy of Ultrasound Assessment of Diaphragmatic Function in Guiding Weaning From Mechanical Ventilation in Critically Ill Patients With Abdominal Sepsis
Brief Title: Diaphragm Ultrasound in Weaning From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Prinicpal investigator, Lecturer of anesthesia and critical care medicine, Cairo University
Other Study IDs: N-16-2017
Record Dates: First submitted 2017-03-15; First posted 2017-03-29 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Sepsis
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the efficacy of ultrasound derived variables in prediction of success of weaning from mechanical ventilation in critically ill patients with abdominal sepsis

DETAILED DESCRIPTION:
Difficult weaning from mechanical ventilation (MV) is a common problem in critically ill patients. Many parameters have been developed to aid weaning from MV such as P/F ratio (PO2/FiO2) and rapid shallow breathing index (respiratory rate/tidal volume); however, sensitivity and specificity for most variables are still variable in literature.

Diaphragmatic dysfunction is a common cause of weaning failure (2) however most of the traditional methods used for evaluation of diaphragmatic function (fluoroscopy, trans-diaphragmatic pressure measurement) are invasive and not available.

Ultrasound assessment of diaphragmatic function has been developed recently providing an easy and safe method for evaluation of diaphragmatic excursion and thickening. In this study we will evaluate the ability of the diaphragmatic function to predict weaning success in patients with abdominal sepsis.

After weaning, patients will be divided into two groups; group of successful weaning (group S) and group with failed weaning (group F) both groups will be compared as regards all clinical, laboratory, and ultrasonographic parameters recorded before weaning, further analysis will be done for patients with repeated trials of weaning (more than one trial or more than one week MV) and those with simple weaning (first time for weaning).

A 7-10 Mega Hertz linear ultrasound probe (Mindray machine) set to B mode, the diaphragm will be visualized by placing the transducer perpendicular to the chest wall, in the eighth or ninth intercostal space, between the anterior axillary and the midaxillary lines, to observe the zone of apposition of the muscle 0.5 to 2 cm below the costophrenic sinus.

The diaphragm thickness will be measured from the middle of the pleural line to the middle of the peritoneal line. Then, the diaphragmatic fraction thickening (DTF) will be calculated as percentage Diaphragmatic movement will be measured in all patients with a 3.5 Mega Hertz US probe placed over one of the lower intercostal spaces in the right anterior axillary line for the right diaphragm and the left midaxillary line for the left diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with abdominal sepsis with history of MV for more than 48 hours

Exclusion Criteria:

* Age < 18 years and surgical dressings over the right lower rib cage which would preclude ultrasound examination will be excluded. Also, patients with chest trauma, thoracotomy, diaphragmatic paralysis, diaphragmatic dysfunction, diaphragmatic injury, diaphragmatic surgery and patients with neuromuscular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with abdominal sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | five minutes before spontaneous breathing trial
  (calculated as maximum thickness - minimum thickness / maximum thickness)

SECONDARY OUTCOMES:
Diaphragmatic excursion | five minutes before spontaneous breathing trial and five minutes before patient extubation
  (measured in millimeters)
Rapid shallow breathing index (RSBI) | five minutes before spontaneous breathing trial
  Respiratory rate/tidal volume in litres
Arterial blood gases | five minutes before spontaneous breathing trial and five minutes before patient extubation
  Partial oxygen pressure and Partial carbon dioxide pressure
Number of weaning trials | during the last 7 days
  number of weaning trials before this trial
Heart rate | five minutes before spontaneous breathing trial and five minutes before patient extubation
  the patient heart rate measured as beat.minute
Arterial blood pressure | five minutes before spontaneous breathing trial and five minutes before patient extubation
  systolic and diastolic blood pressure measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eltrabili HH, Hasanin AM, Soliman MS, Lotfy AM, Hamimy WI, Mukhtar AM. Evaluation of Diaphragmatic Ultrasound Indices as Predictors of Successful Liberation From Mechanical Ventilation in Subjects With Abdominal Sepsis. Respir Care. 2019 May;64(5):564-569. doi: 10.4187/respcare.06391. Epub 2019 Jan 22. PMID 30670667